CLINICAL TRIAL: NCT04586387
Title: The Effect of Brain Anatomy on the Efficacy of Brain Stimulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM20018505
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: transcranial magnetic stimulation; non-invasive brain stimulation; magnetic resonance imaging

STUDY DESIGN:
Masking Description: Participants will not be able to tell the difference if they are being given active vs sham stimulation but will receive both.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Brain stimulation over bicep muscle than finger (FDI) muscle. (Experimental): Brain stimulation will occur over two sessions. Both sessions will occur with sham stimulation then active stimulation. There will be a 3 day rest period between the two muscle groups.
  Interventions: Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over bicep muscle; Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over finger muscle
- Brain stimulation over than finger (FDI) muscle than bicep muscle. (Experimental): Brain stimulation will occur over two sessions. Both sessions will occur with sham stimulation then active stimulation. There will be a 3 day rest period between the two muscle groups.
  Interventions: Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over bicep muscle; Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over finger muscle

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over bicep muscle — repetitive non-invasive brain stimulation protocol which feels like many quick, light taps on your head
Device: intermittent theta burst stimulation (iTBS) with sham and then active stimulation over finger muscle — repetitive non-invasive brain stimulation protocol which feels like many quick, light taps on your head

SUMMARY:
The purpose of this research study is to determine whether brain anatomy impacts the efficacy of transcranial magnetic stimulation (TMS) which is a form of non-invasive brain stimulation. TMS is used to stimulate different areas of the brain and it is well tolerated and generally a safe procedure. It has been studied by researchers for 20 plus years. This brain stimulation device and technique used in this study is an investigational device that has not been approved by the U.S. FDA for treating any muscle or nerve problems. A copy of the device brochure can be found at: https://www.magstim.com/product/rapid-family/

ELIGIBILITY:
Inclusion Criteria:

* nonimpaired individuals
* free of contraindications for MRI and TMS

Exclusion Criteria:

* musculoskeletal injury of the arm
* neurologic deficit affecting motor or sensory function
* concurrent severe medical illness
* diagnosis of SARS-CoV2, or symptoms consistent with COVID-19, or close contact with someone with SARS-CoV2 in the past 3 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Peterson, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total enrollment was 12 with all participants receiving both interventions
Groups:
- Brain Stimulation: Biceps Then FDI; Brain Stimulation: FDI Then Biceps: Brain stimulation
Period: Overall Study
Arm/Group | Brain Stimulation: Biceps Then FDI | Brain Stimulation: FDI Then Biceps
Started | 6 | 6
Sham Stimulation (Will occur over biceps or FDI depending on which area is being stimulated first) | 6 | 6
Active Stimulation (Will occur over biceps or FDI depending on which area is being stimulated first) | 6 | 6
3 Day Rest | 6 | 6
Sham Stimulation (Will occur over biceps or FDI depending on which area is being stimulated second) | 6 | 6
Active Stimulation (Will occur over biceps or FDI depending on which area is being stimulated second) | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This combines both groups.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
Normalized corticomotor excitability [Mean (Standard Deviation); unit: Unitless (a normalized value)] — MEP amplitudes were calculated from the motor target EMG data of each session. Root mean square (RMS) amplitude was calculated for the evoked response over 50ms window (12-62ms post TMS pulse), & for 50ms window prior to the TMS pulse (pre-stimulus). Instances where pre-stimulus RMS exceeded evoked response RMS were excluded. MEPs then normalized & presented as a percentage of the MVC EMG. Normalized MEPs (nMEPs) served as measure of corticomotor excitability, with average of nMEPs collected prior to iTBS serving as baseline. A higher value of nMEP represents greater corticomotor excitability.
  Unitless (a normalized value) | 0.3891 (0.314)

OUTCOME MEASURES:

1. Primary Outcome: Change in Corticomotor Excitability With Active Stimulation on Bicep Muscle
Description: The amplitude the motor evoked potentials (MEPS) will be used to determine level of corticomotor excitability
Time Frame: approximately 7 days
Population: nonimpaired
Measure: Mean (Standard Deviation); unit: percentage of Mwave
Groups:
- All Study Participants: Both study groups
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
percentage of Mwave | 6.9 (3.4)

2. Primary Outcome: Change in Corticomotor Excitability With Sham Stimulation on Bicep Muscle
Description: The amplitude the motor evoked potentials (MEPS) will be used to determine level of corticomotor excitability
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: percentage of Mwave
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
percentage of Mwave | 4.4 (3.2)

3. Primary Outcome: Change in Corticomotor Excitability With Active Stimulation on Finger Muscle
Description: The amplitude the motor evoked potentials (MEPS) will be used to determine level of corticomotor excitability
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: percentage of Mwave
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
percentage of Mwave | 8.6 (5.4)

4. Primary Outcome: Change in Corticomotor Excitability With Sham Stimulation on Finger Muscle
Description: The amplitude the motor evoked potentials (MEPS) will be used to determine level of corticomotor excitability
Time Frame: approximately 7 days
Measure: Mean (Standard Deviation); unit: percentage of Mwave
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
percentage of Mwave | 4.2 (3.1)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Brain Stimulation: intermittent theta burst stimulation (iTBS): repetitive non-invasive brain stimulation protocol which feels like many quick, light taps on your head
Arm/Group | Brain Stimulation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04586387/Prot_SAP_000.pdf